CLINICAL TRIAL: NCT04582240
Title: Full Data BDI Digestif RSCM
Brief Title: Bile Duct Injury Digestif
Status: Completed | Type: Observational
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Vania Myralda Giamour Marbun, Staff of Digestive Division - General Surgery Department, Dr Cipto Mangunkusumo General Hospital
Other Study IDs: BDITJML
Record Dates: First submitted 2020-10-03; First posted 2020-10-09 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Surgery; Biliary Disease; Bile Duct Injury; Sepsis; Jaundice, Obstructive
MeSH Terms: conditions — Gallbladder Diseases; Sepsis; Jaundice, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Data accumulated from medical record collected from January 2008 until December 2018

ELIGIBILITY:
Inclusion Criteria:

* adult patients with extrahepatic bile duct injury managed by digestive division of Cipto Mangunkusumo hospital

Exclusion Criteria:

* none

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients who experienced complication after performed cholecystectomy, open or laparoscopy, related to biliary duct
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Management of Post-Cholecystectomy Bile Duct Injuries without Operative Mortality at Jakarta Tertiary Hospital in Indonesia | january 2008 until december 2018
  Mortality Rate of Patients Performed Reconstructive Surgery for the Management of Bile Duct Injury Post-Cholecystectomy

SECONDARY OUTCOMES:
Management of Post-Cholecystectomy Bile Duct Injuries without Operative Mortality at Jakarta Tertiary Hospital in Indonesia | january 2008 until december 2018
  Most Frequent Anatomical Location of Bile Duct Injury Post-Cholecystectomy